CLINICAL TRIAL: NCT05876806
Title: A Phase II, Open-label Study of Dabrafenib Plus Trametinib in Patients With Advanced Solid Tumor Having BRAF V600E Mutation or Clinically Actionable BRAF Gene Alterations
Brief Title: Dabrafenib Plus Trametinib in Patients With Advanced Solid Tumor Having BRAF V600E Mutation or Clinically Actionable BRAF Gene Alterations
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Se Jun Park (Other)
Responsible Party: Sponsor-Investigator, Se Jun Park, Clinical Assistant Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BROAD
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dabrafenib + Trametinib (Experimental): Subjects will receive Dabrafenib 150 mg twice daily orally plus Trametinib 2 mg once daily orally on a continuous basis. A treatment cycle is 28 days in duration. Subjects will continue treatment until an unacceptable toxicity, disease progression, or death occurs.
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib is a 150 mg twice daily capsule administered orally on a continuous basis
Drug: Trametinib — Trametinib is a 2 mg once daily tablet administered orally on a continuous basis.

SUMMARY:
This is a Phase II, open-label, non-randomized, multi-center study of oral Dabrafenib in combination with oral Trametinib in subjects with solid tumors with BRAF V600E mutation or clinically actionable BRAF gene alterations.

DETAILED DESCRIPTION:
Dabrafenib and trametinib combination treatment can offer a therapeutic option for patients with solid cancers harboring specific gene mutations, for whom there are no alternative treatments.

Patients with BRAF V600 mutated advanced solid tumor (excluding BRAF V600E/K mutated malignant melanoma, BRAF V600E mutated non-small cell lung cancer, and BRAF V600E mutated colorectal cancer) or patients with other BRAF gene alterations that are regarded to be druggable by the KOSMOS MTB.

This study is designed to determine the disease control rate (DCR) of oral Dabrafenib in combination with oral Trametinib in subjects with BRAF V600E or clinically actionable BRAF mutated cancers. Only subjects with histologically confirmed advanced disease and no available standard treatment options will be eligible for enrollment. Subjects will undergo screening assessments within 30 days prior to the start of treatment to determine their eligibility for enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria for study entry:

1. Patient who agreed to participate in the KOSMOS-II master observation study
2. 19 years of age or older
3. Patients with BRAF V600 mutated advanced solid tumor (excluding BRAF V600E/K mutated malignant melanoma, BRAF V600E mutated non-small cell lung cancer, and BRAF V600E mutated colorectal cancer)
4. Patients with other BRAF gene alterations that are regarded to be actionable by the KOSMOS MTB
5. Disease progression after ≥ 1-prior line of systemic treatment and no standard treatment option
6. ECOG performance status score 0-2
7. Life expectancy of > 3 months
8. Measurable or evaluable disease according to RECIST version 1.1
9. Ability to take oral medications
10. Adequate bone marrow and organ function
11. Patients who voluntarily decided to participate after understanding this clinical trial, and signed a written informed consent

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from study entry:

1. Prior treatment with a BRAF inhibitor (including, but not limited to, dabrafenib, vemurafenib, encorafenib) or MEK inhibitor (including, but not limited to, trametinib, binimetinib, selumetinib, cobimetinib) or ERK inhibitor (including, but not limited to, ravoxertinib, ulixertinib, CC-90003, MK-8353)
2. History of malignancies with confirmed activating RAS mutation.
3. Hypersensitivity to the active ingredients and additives of investigational product.
4. Presence of any unresolved ≥Grade 2 (per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0) toxicity from previous anti-cancer therapy at the time of enrollment. (Except toxicities which are not clinically significant such as alopecia, skin discoloration, and neuropathy).
5. Any anti-cancer treatment (local treatment, chemotherapy, immunotherapy, targeted therapy) within 2 weeks prior to the start of study treatment.
6. Prior major surgery less than 14 days before enrollment. Any surgery-related AE must have been resolved before enrollment.
7. Prior radiotherapy less than 14 days before enrollment, except for ATC (radiotherapy is not permitted within 7 days before enrollment).
8. Known additional malignancy that is progressing or has required active treatment within the past 3 years. (Patient with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma is potentially eligible).
9. Presence of central nervous system metastases that are symptomatic or untreated or not stable for ≥3 months or requiring corticosteroids.
10. Symptomatic or untreated leptomeningeal or spinal cord compression. Subjects who have been previously treated for these conditions are asymptomatic and currently not taking corticosteroids before enrollment, is permitted.
11. Current evidence of cardiovascular risk including any of the following:

    * Left ventricular ejection fraction (LVEF) below the institutional lower limit of normal
    * QT interval corrected for heart rate using Bazett's formula ≥ 480 msec
    * Clinically significant uncontrolled arrhythmias
    * Moderate valvular thickening documented by echocardiography
    * Presence of intra-cardiac defibrillators
    * Acute coronary syndromes (including myocardial infarction and unstable angina) which required coronary angioplasty or stenting within 6 months before enrollment
    * Congestive heart failure ≥ Class II as defined by New York Heart Association
12. Current evidence or history of retinal vein occlusion
13. Pregnant or lactating women
14. Patients who do not consent to adequate contraception throughout the study period

    * Women of childbearing potential should use effective contraception* until 16 weeks after the last investigational product administration
    * Male patients who have not undergone a vasectomy must consent to the use of appropriate contraception* and are prohibited from providing sperm for up to 16 weeks after administration of the last investigational product * Appropriate contraception: hormonal contraceptives (subcutaneous formulas, injections, oral contraceptives, etc.), intrauterine devices (IUD, Intra Uterine Device or IUS, Intra Uterine System), sterilization by participants or participant's partner (vasectomy, tubal ligation, etc.); Double blocking (a method that uses a combination of blocking methods, such as using a cervical cap or a contraceptive diaphragm with a male condom)
15. Active infection such as hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)

    * For HBsAg is positive, and HBV DNA ≤ LLOQ, enrollment of the subject can be considered.
    * If the patient with chronic hepatitis B who are HBsAg positive and HBV DNA positive has been taking antiviral drugs for more than 3 months, enrollment of the subject can be considered at the investigator's discretion.
    * For IgG anti-HBc is positive (a history of HBV infection) and HBV DNA ≤ LLOQ, enrollment of the subject can be considered.
    * For Anti-HCV Ab is positive, and HCV RNA ≤ LLOQ, enrollment of the subject can be considered.
16. Acute/chronic medical or psychiatric abnormalities
17. The investigator judges that it is not appropriate to participate in this study for else reasons.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | From study treatment start date until first documented complete response, partial response or stable disease, assessed up to 36 months
  Disease control Rate (DCR) is defined as the proportion of subjects with objective evidence of complete response (CR), partial response (PR), or stable disease (SD).

SECONDARY OUTCOMES:
Overall Survival (OS) | From study treatment start date until date of of death from any cause, assessed up to 36 months
  Overall Survival (OS) is defined as the time from first dose until death due to any cause.
Progression Free Survival (PFS) | From study treatment start date until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 36 months
  Progression Free Survival (PFS) is defined as the interval between the first dose of study treatment and earlier date of first radiologically documented progression or death due to any cause.
Objective Response Rate (ORR) | From study treatment start date until first documented complete response or partial response, assessed up to 36 months
  Overall Response Rate (ORR) is defined as the percentage of participants with a confirmed overall response by investigator assessment as defined by the pre-specified response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Se Jun Park, MD, PhD, Principal Investigator — The Catholic University of Korea
Locations (1):
- Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul, South Korea